CLINICAL TRIAL: NCT06548009
Title: Serum Metabolics-based Method for Diagnosing Bile Acid Diarrhoea
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Asger Lund, MD, MD, PhD, University Hospital, Gentofte, Copenhagen
Other Study IDs: BAD-DIVA
Record Dates: First submitted 2024-05-03; First posted 2024-08-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Bile Acid Malabsorption; Bile Acid Diarrhea
Keywords: bile acid; diarrhea; diagnostics
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SeHCAT confirmed bile acid diarrhea: Patients referred to a SeHCAT scan due to suspected bile acid diarrhea, who afterwards turned out to be suffering from SeHCAT confirmed bile acid diarrhea
  Interventions: Diagnostic Test: Metabolomics and other blood samples
- SeHCAT negative patients: Patients referred to a SeHCAT scan due to suspected bile acid diarrhea, who afterwards turned out to be SeHCAT negative
  Interventions: Diagnostic Test: Metabolomics and other blood samples

INTERVENTIONS:
Diagnostic Test: Metabolomics and other blood samples — Blood samples taken with the objective of identifying a diagnostic test

SUMMARY:
Bile acid diarrhoea (BAD) is a common yet under-diagnosed and under-recognised disease. The primary symptoms are watery diarrhoea with high frequency of unpredictable bowel movements,urgency and faecal incontinence making BAD a debilitating condition. One of the challenges of BAD is the lack of a readily available and accurate diagnostic test.

The aim of this study is to validate a BAD diagnostic score (BDS) based on metabolomics.

DETAILED DESCRIPTION:
Bile acid diarrhoea (BAD) is a common yet under-diagnosed and under-recognised disease. The primary symptoms are watery diarrhoea with high frequency of unpredictable bowel movements,urgency and faecal incontinence making BAD a debilitating condition. The pathophysiology of BAD involves spill-over of bile acids to the colon where bile acids irritate the colonic mucosa and cause osmotic-induced fluid secretion. The aetiology of BAD can be either idiopathic (termed primary BAD or type 2 BAD) or the disease can develop secondary to ileal dysfunction (due to, e.g., intestinal surgery or Chron's disease, termed type 1 BAD) or other conditions interfering with ileal absorption (due to, e.g., cholecystectomy or radiation therapy, termed type 3 BAD).

Irritable bowel syndrome (IBS) with predominant diarrhoea is a common condition in the general population (prevalence of around 4%) and emerging data suggest that around 1/3 suffering from this condition in fact have BAD. Many of these patients remains undiagnosed and thus,inappropriately treated or even untreated. A major reason for this is challenges associated with diagnosing BAD. Several diagnostic modalities have been suggested including 14C-glycocholate breath test, stool test and assessment of 48-hour faecal bile acid output. These tests are cumbersome, time-consuming, and not widely available. The 75selenium homocholic acid taurine (SeHCAT) test is considered the gold standard for the diagnosis of BAD. It measures, via a standard gamma camera, the 7-day retention of a taurine-conjugated bile acid analogue labelled with the gamma-emitter 75selenium. This test provides a quantitative assessment to estimate the severity of BAD, but there is no general agreement regarding its cut-off value and the test is not widely available or even approved for clinical use in many countries outside Europe, including the USA. Furthermore, the SeHCAT test is cumbersome due to its dependence on two visits to the clinic exactly seven days apart, it is expensive, and involves radioactive exposure to the patient. Given the limited availability and the challenges associated with the abovementioned tests, excluding BAD is unfortunately not within current routine investigational algorithms for diarrhoea-predominant IBS, Crohn's disease, or gastrointestinal cancers. In many cases, BAD diagnosis is considered after therapeutic trial using bile acid sequestrants. However, these agents are expensive, often ineffective and/or associated with gastrointestinal side effects in patients with established BAD why their potential as diagnostic tools is limited. Taken together, diagnosing BAD is currently associated with challenges that may preclude relevant treatment of this debilitating condition warranting development of easy and accessible yet safe and effective BAD diagnostics. Recently, the investigators have developed a new BAD diagnostic method based on a single blood sample from the patient. Our approach is based on unbiased, metabolic profiling of serum from BAD patients and carefully matched healthy individuals using comprehensive ultra-high-performance liquid chromatography time-of-flight mass-spectrometry. These comprehensive datasets were subjected to state-of-the-art machine learning and used to build a BAD diagnostic score (BDS) that can distinguish a patient suffering BAD from healthy individuals with high precision (sensitivity of 78% and specificity of 93%). In the present study, the investigators will refine the BDS to distinguish between patients suffering from BAD and patients suffering from other diarrhoeal diseases by using the same methods and data analyses as in the previous project, but in this case applied to serum samples collected from patients referred to diagnostic SeHCAT test, i.e., samples from both test-positive and test-negative patients.

ELIGIBILITY:
Inclusion Criteria:

* SeHCAT referral for suspected bile acid diarrhoea
* Age ≥18 years

Exclusion Criteria:

* Diabetes, except type 2 diabetes
* Nephropathy with estimated glomerular filtration rate <30 min/1.73 m2
* Treatment with medicine that cannot be paused for 12 hours
* Hypothyroidism or hyperthyroidism, if not well regulated
* Active or recent (<6 months since last treatment) malignant disease
* Any treatment or condition requiring acute or subacute medical or surgical intervention
* Any condition considered incompatible with trial participation by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of SeHCAT referred patients for suspected bile acid diarrhoea.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
AUROC curve of the BDS in the validation cohort | 1 year from now
  AUROC curve of the BDS in the validation cohort

SECONDARY OUTCOMES:
AUROC curve of BDS in patients with each of the three subtypes of BAD | 1 year from now
AUROC curve of BDS in the discovery cohort (see 8.2 Data analysis) | 1 year from now
Correlation of SeHCAT test result with severity of BAD symptoms | 1 year from now
Correlation of BDS test results with number of stools per day | 1 year from now
Biomarkers for BAD: C4 and FGF19 | 1 year from now

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Bispebjerg and Frederiksberg Hospital, Copenhagen
  - Herlev Gentofte Hospital, Hellerup
  - Hillerød Hospital, Hillerød

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewinska M, Karhus ML, Ellegaard AG, Romero-Gomez M, Macias RIR, Andersen JB, Knop FK. Serum lipidome unravels a diagnostic potential in bile acid diarrhoea. Gut. 2023 Sep;72(9):1698-1708. doi: 10.1136/gutjnl-2022-329213. Epub 2023 Apr 18. PMID 37072179